CLINICAL TRIAL: NCT02130063
Title: A Phase III, Randomised, Open-Label, Comparative Study of Intravenous Iron Isomaltoside 1000 (Monofer®) and Iron Sucrose in Subjects With Iron Deficiency Anaemia and Who Are Intolerant or Unresponsive to Oral Iron Therapy or Who Need Iron Rapidly (PROVIDE)
Brief Title: IDA-01 A Randomised, Open-Label, Comparative Study of Intravenous Iron Isomaltoside 1000 (Monofer®) and Iron Sucrose
Acronym: Provide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry); ClinStar, LLC (Industry); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IDA-01
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2015-08

CONDITIONS: Iron Deficiency Anaemia
Keywords: IDA; Iron deficiency; iron deficiency anaemia and who are intolerant or unresponsive to oral iron therapy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — iron isomaltoside 1000; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron isomaltoside 1000 (Monofer®) (Experimental): iron isomaltoside 1000 (Monofer®)
  Interventions: Drug: iron isomaltoside 1000 (Monofer®)
- iron sucrose (Venofer®) (Active Comparator): iron sucrose (Venofer®)
  Interventions: Drug: iron sucrose (Venofer®)

INTERVENTIONS:
Drug: iron isomaltoside 1000 (Monofer®)
  Arms: iron isomaltoside 1000 (Monofer®)
Drug: iron sucrose (Venofer®)
  Arms: iron sucrose (Venofer®)

SUMMARY:
The purpose of the trial is to evaluate and compare the effect of iron isomaltoside 1000 to iron sucrose in its ability to increase haemoglobin (Hb) in subjects with IDA when oral iron preparations are ineffective or cannot be used or where there is a clinical need to deliver iron rapidly.

DETAILED DESCRIPTION:
IDA is highly prevalent in subjects with gastrointestinal diseases and cancer, menstruating or pregnant women, and subjects who have undergone bariatric procedure. IDA can have a substantial medical and quality of life (QoL) burden on the subjects and the treatment of these subjects includes controlling the bleeding and replenishing lost iron. Oral iron administration is often used in the clinical practice at many clinics; however, oral iron may not be tolerated by all subjects. Hence, there is a need for an alternative iron treatment in subjects, who do not tolerate oral iron.

This study is planned to compare the efficacy and safety of iron isomaltoside 1000 with another parenteral iron preparation (iron sucrose) in subjects with IDA and who are intolerant or unresponsive to oral iron therapy or who need iron rapidly.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women > 18 years having IDA caused by different aetiologies such as abnormal uterine bleeding, gastrointestinal diseases, cancer, bariatric procedures (gastric bypass operations), and other conditions leading to significant blood loss and with a documented history of intolerance or unresponsiveness to oral iron therapy for at least one month prior to study enrollment or where there at investigators judgment is a clinical need to deliver iron rapidly
2. Hb < 11 g/dL
3. TSAT < 20 %
4. S-ferritin < 100 ng/mL
5. Willingness to participate and signing the informed consent form

Exclusion Criteria:

1. Anaemia predominantly caused by factors other than IDA (e.g. anaemia with untreated vitamin B12 or folate deficiency, haemolytic anaemia)
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
3. Decompensated liver cirrhosis or active hepatitis (ALAT > 3 times upper limit of normal)
4. Active acute or chronic infections (assessed by clinical judgement supplied with white blood cells (WBC) and C-reactive protein (CRP))
5. Body weight < 50 kg
6. Rheumatoid arthritis with symptoms or signs of active inflammation
7. Pregnant or nursing women. In order to avoid pregnancy, women have to be surgically sterile or use adequate contraception (e.g. intrauterine devices, hormonal contraceptives, or double barrier method) during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product
8. History of multiple allergies
9. Known hypersensitivity to parenteral iron or any excipients in the investigational drug products
10. Erythropoietin treatment within 8 weeks prior to the screening visit
11. Other iron treatment or blood transfusion within 4 weeks prior to the screening visit
12. Planned elective surgery during the study
13. Participation in any other clinical study within 3 months prior to the screening
14. Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study, e.g. uncontrolled hypertension, unstable ischaemic heart disease, or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmington, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
Started | 342 | 169
Completed | 317 | 152
Not Completed | 25 | 17

BASELINE CHARACTERISTICS:
Population: FAS (N = 491): The FAS consisted of all subjects who were randomised, received at least one dose of the trial drug, and had at least one post-baseline Hb assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®) | Total
Number analyzed (Participants) | 342 | 169 | 511
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (15.8) | 46.8 (14.9) | 48.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309 | 154 | 463
  Male | 33 | 15 | 48
Region of Enrollment [Number; unit: participants]
  United States | 342 | 169 | 511

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Haemoglobin (Hb) Increase of ≥ 2 g/dL From Baseline at Any Time From Week 1 to Week 5
Description: The primary efficacy endpoint of the trial was the count of subjects with an Hb increase of ≥ 2 g/dL from baseline at any time from week 1 to week 5. 'Any time' implied that if the endpoint was met at a time-point prior to or at week 5, the effect (increase of ≥ 2 g/dL) did not have to be maintained throughout the trial in order for a subject to be a responder.
  Number of responders (i.e. a subject with increase in Hb ≥ 2 g/dL from baseline at any time from week 1 to week 5) and percentages according to number of subjects in the analysis set were summarised.
Time Frame: From baseline to week 5
Population: Full analysis set (FAS) (N = 491): The FAS consisted of all subjects who were randomised, received at least one dose of the trial drug, and had at least one post-baseline Hb assessment.
Measure: Number; unit: participants
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
Number analyzed (Participants) | 330 | 161
participants | 226 | 83

2. Secondary Outcome: Change in Hb Concentration
Time Frame: From baseline to week 2, 4 and 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
Number analyzed (Participants) | 330 | 161
g/dL
  Week 2 | 1.56 (1.03) | 0.87 (0.90)
  Week 4 | 2.35 (1.32) | 1.74 (1.17)
  Week 5 | 2.52 (1.41) | 2.05 (1.27)

3. Secondary Outcome: Change in Serum (s)-Ferritin Concentration
Time Frame: From baseline to week 1, 2, 4, and 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
Number analyzed (Participants) | 330 | 161
ng/mL
  Week 1 | 431.2 (221.4) | 86.9 (84.8)
  Week 2 | 516.6 (268.1) | 126.2 (87.2)
  Week 4 | 285.3 (205.2) | 195.0 (126.2)
  Week 5 | 241.2 (209.3) | 185.7 (166.8)

4. Secondary Outcome: Change in Transferrin Saturation (TSAT)
Time Frame: From baseline to week 1, 2, 4, and 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
Number analyzed (Participants) | 330 | 161
percent
  Week 1 | 15.7 (9.6) | 3.3 (8.1)
  Week 2 | 17.9 (9.8) | 5.7 (6.8)
  Week 4 | 16.3 (9.0) | 11.5 (9.5)
  Week 5 | 15.6 (8.6) | 11.8 (9.5)

ADVERSE EVENTS:
Time Frame: From screening until week 5
Description: The nature of the event will be described in precise, standard medical terminology. If known, a specific diagnosis was stated. Furthermore the Investigator described an AE regarding seriousness, severity, relatedness, and outcome.
  It is only the subjects that received treatment that is included in the safety analysis. Of the 342 enrolled subjects in the Monofer arm only 333 was treated. Of the 169 subjects enrolled in the Venofer arm 168 was treated.
Arm/Group | Iron Isomaltoside 1000 (Monofer®) | Iron Sucrose (Venofer®)
All-Cause Mortality (participants affected / at risk) | 1/333 | 0/168
Serious Adverse Events (participants affected / at risk) | 11/333 | 6/168
Other Adverse Events (participants affected / at risk) | 100/333 | 54/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (Monofer®) (N=333) | Iron Sucrose (Venofer®) (N=168)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stent malfunction (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (Monofer®) (N=333) | Iron Sucrose (Venofer®) (N=168)
Nausea (Gastrointestinal disorders) | 17 (19) | 7 (8)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (6)
Urinary tract infection (Infections and infestations) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (3)
Dizziness (Nervous system disorders) | 9 (10) | 4 (5)
Headache (Nervous system disorders) | 18 (21) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 14 (18) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (7)
Dysgeusia (Nervous system disorders) | 2 (2) | 5 (10)
Fatique (General disorders) | 4 (4) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No